CLINICAL TRIAL: NCT05535556
Title: Comparison of the Electric Plasma Surgical Tool "PlasmaBlade" for Replacement of the Deep Brain Stimulation (DBS) Devices With Conventional Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2021-0063
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia; Epilepsy
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The deep brain stimulation is surgical technique used for the Parkinson's disease, essential tremor, dystonia, epilepsy, and psychiatric diseases. A pulse generator or battery (implanted pulse generator, IPG) is a need for replacement every few years. In general, electric cautery(BOVIE), which is commonly used in surgery, cannot be used when the deep brain stimulation machine is inserted, so conventional tools such as scissors and knives are used for replacement surgery. However, in the process, damage to the machine may be inflicted by knives, scissors, etc., and in the worst case, the machine may be unusable, resulting in financial and human consumption.

Plasma Blade is currently used for tissue incision and coagulation in Korea, and is the only insurance-recognized tool in Korea for the replacement surgery of a cardiovascular implantable electronic device (CIED). The deep brain stimulation machine has a structure very similar to that of the heart electronics. In addition, the plasma blade was used to replace the deep brain stimulation machine overseas.The safety is reported in the surgery, so the plasma blade deep brain stimulation machine has been replaced in Korea. The investigators would like to check the safety and effectiveness for use in surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 19
* Those who voluntarily agree to participate in this clinical trial and are willing to comply with the clinical trial protocol
* Persons who have previously undergone deep brain stimulation for Parkinson's disease, essential tremor, dystonia, epilepsy, etc.
* Those who need replacement of deep brain stimulation machine

Exclusion Criteria:

* Those who cannot be under general anesthesia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For those who need to replace the deep brain stimulation machine, and those who have given voluntary consent
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-07-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
Complications occurred during surgery | Immediately after surgery
  Evaluate mechanical damage to the DBS machine immediately after surgery

SECONDARY OUTCOMES:
Surgical time | Intraoperative
  Check the time required for surgery
The occurrence of wound-related complications | The 1 day after surgery, 3 weeks after surgery, 6 months after surgery
  the occurrence of short-term/long-term complications (hematoma, infection, wound spread, and changes in mechanical resistance values) the 1 day after surgery, 3 weeks after surgery, and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Chang, Principal Investigator — Department of Neurosurgery, Brain Research Institute, Yonsei University College of Medicine, Seoul, South Korea
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No